CLINICAL TRIAL: NCT01919060
Title: Acute Non-mechanical Lower Digestive Tract Disorders Should Distinguish Whether Colonic Lesions or Not in Critically Ill Patients
Status: Completed | Type: Observational
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: Principal Investigator, Gao Tao, Nanjing university, Nanjing PLA General Hospital
Other Study IDs: 2007NLY099
Record Dates: First submitted 2013-08-06; First posted 2013-08-08 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2007-01

CONDITIONS: Critical Care Patient; Lower Digestive Tract Disorder;; Colon Lesions;

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- lesions in colon
- lesions in extra-colon

SUMMARY:
The purpose of the study is to investigate acute non-mechanical lower digestive tract disorders should distinguish whether colonic lesions or not in critically ill patients

DETAILED DESCRIPTION:
The study was approved by the ethics committee of Jinling hospital and the medical school of nanjing university. This prospective study was performed at a surgical intensive care unit (SICU), which contain 39 beds, of general surgical departement of Jinling hospital, affiliated hospital of medical school of nanjing university. Written informed consents were obtained from the patients or their next of kin.

Critical patients aging from 18 to 80 years old diagnosed with acute lower gastrointestinal dysfunction were recrutied to the study. The two following criterias should met for the diagnosis of acute lower gastrointestinal dysfunction: 1. enteral nutrition intolerance not due to upper gastriointestinal obstruction; 2. Colonic distension: colonic diameter >6 cm or ileocecus diameter >9 cm under the view of computed tomography or abdomial X ray. Enteral nutrition intolerance was defined as enteral feeding < 50% caculated needs or no feeding for three days.

Patients with following conditions were excluded: mechanical intestinal obstruction (including tomor, stercoral obstruction etc); gastrointestinal hemorrhage within 72 hours; history of inflammatory bowel disease (ulcerative colitis or crohn's disease) or radiation enteritis; pregnancy; having the contradiction of proserine administration.

Data on demagraphy, diagnosis, treatment as well as APACHE Ⅱ and SOFA score within 24 hs of admission were recorded. The included patients were examined by contrast-enhanced abdominal CT, and were devided into two groups, colon oriented group and non-colon oriented group, independently by 2 professionals combining the history and CT results. Non-colon oriented group should met one of the two following crieria: 1. with a history of nerves damage which affect colon movement (colon(-innervating) nerves damage) (such as pevic or retroperitoneal operation, spine injury, cerebral lesion), and non- or mild edema of colonic wall presented on abdominal CT; 2. without a history of colon(-innervating) nerves damage, whereas no obvious change can be seen on CT scan. The others were clarified as colon-oriented group (namely, with a history of colon(-innervating) nerves damage, moderate or more severe edema; without a history of colon(-innervating) nerves damage, whereas mild or sever edema presented ).

All the patients diagnosed with acute lower gastrointestinal dysfunction were treated according to the protocol depicted in figure 1.

Conservative treatment: firstly, hydro-electrolyte and thyroid function were assessed, and corrected if abnormal. Maintain the blood glucose at the normal level. Patients proning to be diagnosed with sepsis were adminstered antibiotics empirically, and adjusted to more targeted antibiotics according to the ensuing result of blood culture and drug sensitive test. Patients were subject to fasting, gastrointestinal decompression via stomach and anal tube. Gastric residual volume (GRV) was assessed per diem. Pharmaceuticals impacting bowel movement were suspended as far as possible, such as opiate, anticholinergic drugs, and calcium channel blockers (CCB). Intravenous administration of proserine was considered if cecum diameter > 10 cm after the treatement described above and show no signs of ameliaration in 24 h.

Colonoscopic decompression: colonoscopic decompression was applied when obvious cecum distension existed (diameter > 10) more than 3 days, and no signs of improvement gained after 24-48 hs of conservative treatment or contradiction of proserine existed. Colonoscopic decompression was performed by 2 experienced endoscopic physicians at the bedside or in the endoscope room.

Surgical intervention: surgery was indicated when colonic diatension lasted more than 6 days, or obvious cecal distention (diameter > 10 cm) continued after 48-72 hs of conservative management and colonoscopic decompression ???or with contradiction of colonoscopy. ileostomy was performed under epidural or local anesthesia by a team of experienced surgeons. If the patients had colonic necrosis or perforation, ileostomy was superseded by colectomy under general anesthesia.

In the SICU, bladder pressure was measured everaday to reflect intraabdominal pressure. And patients received CT examination at day 1, day 3, day 5 and every eusing week, other than additional illness-required CT. The measurement of colonic or cecum diameter, and assessment of intestional eddema, ischemia and perforation were performed by two trained fellows to record the recovery time. Criteria for colonic recovery were as follows: 1.enteral nutrition reached or surpass 50% of targeted needs more than 3 days; 2. Restoration of normal aerofluxus and defecation; 3. Significant improvent of colonic distension or colonic wall was shown on abdominal CT (colonic diameter < 6 cm or cecum diameter < 9 cm).

Recurrence was defined as, patients rediagnosed with acute lower gastrointestional dysfunction within 72 hrs of recovery after a certain treatment(s).

ELIGIBILITY:
Inclusion Criteria:

1. Critical patients aging from 18 to 80 years old diagnosed with acute lower gastrointestinal dysfunction
2. enteral nutrition intolerance not due to upper gastriointestinal obstruction
3. Colonic distension: colonic diameter >6 cm or ileocecus diameter >9 cm under the view of computed tomography or abdomial X ray. Enteral nutrition intolerance was defined as enteral feeding < 50% caculated needs or no feeding for three days -

Exclusion Criteria:

mechanical intestinal obstruction (including tomor, stercoral obstruction etc); gastrointestinal hemorrhage within 72 hours; history of inflammatory bowel disease (ulcerative colitis or crohn's disease) or radiation enteritis; pregnancy; having the contradiction of proserine administration. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was approved by the ethics committee of Jinling hospital and the medical school of nanjing university. This prospective study was performed at a surgical intensive care unit (SICU), which contain 39 beds, of general surgical departement of Jinling hospital, affiliated hospital of medical school of nanjing university. Written informed consents were obtained from the patients or their next of kin. Critical patients aging from 18 to 80 years old diagnosed with acute lower gastrointestinal dysfunction were recrutied to the study.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2007-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 28

SECONDARY OUTCOMES:
Organ failure or dysfunction | 28day

OTHER OUTCOMES:
colonic diameter | 7day